CLINICAL TRIAL: NCT04957043
Title: Application of 3D Fast Spin-echo Sequence (3D-Matrix) Optimized by Compressed Sensing Technology in Knee Joint Sports Injury
Brief Title: Application of 3D-Matrix in Knee Joint Sports Injury
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018017
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
3 d scan sequence can realize continuous thin layer scanning, the thinnest layer thickness of 0.5 mm, to reduce the effects of partial volume effect and improve the spatial resolution image, the other 3 d sequence can according to need to multiplanar reconstruction based on the original image, the image of the watch is no longer limited to a fixed plane, and can avoid repeated scanning, reducing overall inspection time. Initially, 3D MRI uses gradient echo sequences (3D-GRE). Although the scan time of 3D-GRE is acceptable and has a high spatial resolution, the contrast between tissues is poor. In recent years, is voxel 3D fast spin-echo sequence (3D-FSE) has become an alternative 3D scanning sequence. Compared with the 3D-GRE sequence, 3D-FSE has better-intertissued contrast. However, there are still some problems in the application of 3D sequence in clinical practice. On the one hand, although 3D sequence reduces the overall scanning time, it increases the single scanning time, so it is easy to produce motion artifacts. On the other hand, although many studies have demonstrated the diagnostic efficacy of 3D sequences in the diagnosis of common intraarticular structural injuries, especially in the diagnosis of knee cartilage injuries, the diagnostic value of 3D sequences is comparable to that of conventional 2D-FSE sequences, but the evidence on whether 3D sequences can replace 2D sequences is still insufficient.

Recently, a new fast signal acquisition technology -- Compressed Sensing (Compressed Sensing) technology has been gradually applied to many kinds of MRI sequences, and its application in 3D sequences can greatly shorten the single scan time. In this study, Modulated Flip Angle Technique in Refocused Imaging with Extended Echo was applied by United Imaging Co., Ltd. (Compressed Sensing) Train, 3D-Matrix), which is a fast self-selected echo sequence based on variable turn Angle technology, and its single scan time can be shortened to 5 minutes. 3 d sequence to more systematic evaluation on sports injury of knee joint application value, the investigators will study from within the bony structure of knee joint injury, joint structure damage and injury of the surrounding support structure aspects to discuss the diagnosis effect, and with arthroscopy for the gold standard to evaluate the accuracy of the 3 d structure within the sequence in the diagnosis of knee joint injury.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is the most important non-invasive examination method for the diagnosis of knee joint sports injury. 2D-FSE sequence is usually used for axial, sagittal and coronal scanning in MR examination of the knee joint. The sequence has good tissue contrast and spatial resolution. However, there are still some problems with 2D-FSE sequences. For example, the scanning layer thickness is usually up to 3-5mm, and there is a certain layer spacing, resulting in partial volume effect. In addition, in order to obtain images with different azimuths, the same sequence needs to be scanned for many times, which increases the overall inspection time.

3 d scan sequence can realize continuous thin layer scanning, the most thin layer thickness of 0.5 mm , so as to reduce the effects of partial volume effect and improve the spatial resolution image, the other 3 d sequence can be on the basis of the original image according to need multiplanar reconstruction, make the observation of the image is no longer limited to the fixed plane, and can avoid repeated scanning, reducing overall inspection time. Initially, 3D MRI uses gradient echo sequences (3D-GRE). Although the scan time of 3D-GRE is acceptable and has high spatial resolution, the contrast between tissues is poor. In recent years, the isosvoxel 3D fast spin echo sequence (3D-FSE) has become an alternative 3D scanning sequence. Compared with 3D-GRE sequence, 3D-FSE has better intertissue contrast . However, there are still some problems in the application of 3D sequences in clinical practice. On the one hand, although 3D sequences reduce the overall scanning time, the single scanning time increases. At present, the scanning time in most studies is generally 6-10 minutes , so motion artifacts are easily generated. On the other hand, although many studies have proved the diagnostic efficacy of 3D sequence in the diagnosis of common intraarticular structural injuries , especially the diagnostic value of 3D sequence in the diagnosis of knee cartilage injuries is equivalent to that of conventional 2D-FSE sequence, there is insufficient evidence on whether 3D sequence can replace 2D sequence .

Recently, a new fast signal acquisition technology -- Compressed Sensing (Compressed Sensing) technology has been gradually applied to a variety of MRI sequences , and its application in 3D sequences can greatly shorten the single scan time. In this study, Modulated Flip Angle Technique in Refocused Imaging with Extended Echo was applied by United Imaging Co., Ltd. (Compressed Sensing) Train, 3D-Matrix), which is a fast self-selected echo sequence based on variable turn Angle technology, and its single scan time can be shortened to 5 minutes. 3 d sequence in order to more systematic evaluation on sports injury of knee joint application value, the investigators will study from within the bony structure of knee joint injury, joint structure damage and injury of the surrounding support structure aspects to discuss the diagnosis effect, and with arthroscopy for gold standard to evaluate the accuracy of the 3 d structure within the sequence in the diagnosis of knee joint injury.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clear history of knee injury, clinically suspected knee injury, need MRI examination;
2. Arthroscopy or treatment is planned.

Exclusion Criteria:

1. Patients with the following diseases: rheumatoid arthritis, septic arthritis, tumor, anterior cruciate ligament mucinous degeneration, and articular fibrosis;
2. Previous history of knee surgery;
3. MRI contraindication: patients with metal in body (pacemaker, prosthetic eye, metal implant), pregnancy or claustrophobia;
4. Arthroscopy was not performed after MRI examination for various reasons;
5. The time interval between MRI examination and arthroscopy was more than 2 months.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: About 150 inpatients planned to undergo MRI examination of knee joint
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the image quality of knee joint imaging with 3D-Matrix sequence | 2018-2019
  Evaluate the image quality of knee joint imaging with 3D-Matrix sequence
Evaluate the image accuracy of knee joint imaging with 3D-Matrix sequence | 2018-2019
  Using arthroscopy as the gold standard, the accuracy of 3D-Matrix and conventional 2D-FSE sequences in the diagnosis of anterior cruciate ligament (ACL), meniscus and articular cartilage injuries was compared.

CONTACTS AND LOCATIONS:
Overall Officials: huishu yuan, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China